CLINICAL TRIAL: NCT04793958
Title: A Randomized Phase 3 Study of MRTX849 in Combination With Cetuximab Versus Chemotherapy in Patients With Advanced Colorectal Cancer With KRAS G12C Mutation With Disease Progression On or After Standard First-Line Therapy
Brief Title: Phase 3 Study of MRTX849 With Cetuximab vs Chemotherapy in Patients With Advanced Colorectal Cancer With KRAS G12C Mutation (KRYSTAL-10)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0006; KRYSTAL-10 (Other: Mirati Therapeutics); CA239-0006 (Other: Bristol-Myers Squibb Protocol ID); 849-010 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2021-03-02; First posted 2021-03-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Advanced Colorectal Cancer; Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Colorectal Cancer Trial; Colorectal Carcinoma; Rectal Cancer; Colon Cancer; KRAS; KRAS G12C; RAS; Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — adagrasib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRTX849 + Cetuximab (Experimental)
  Interventions: Drug: MRTX849; Biological: Cetuximab
- mFOLFOX6 or FOLFIRI (Active Comparator)
  Interventions: Drug: mFOLFOX6 Regimen; Drug: FOLFIRI Regimen

INTERVENTIONS:
Drug: MRTX849 — 28 Day Cycle
  Arms: MRTX849 + Cetuximab
Biological: Cetuximab — 28 Day Cycle
  Other Names: Erbitux
  Arms: MRTX849 + Cetuximab
Drug: mFOLFOX6 Regimen — * Fluorouracil
  * Oxaliplatin
  * Folinic acid
  Arms: mFOLFOX6 or FOLFIRI
Drug: FOLFIRI Regimen — * Fluorouracil
  * Irinotecan
  * Folinic acid
  Arms: mFOLFOX6 or FOLFIRI

SUMMARY:
Study CA239-0006 is an open-label, randomized Phase 3 clinical trial comparing the efficacy of MRTX849 administered in combination with cetuximab versus chemotherapy in the second-line treatment setting in patients with CRC with KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal carcinoma with KRAS G12C mutation in tumor tissue.
* Prior receipt of 1st line treatment in advanced CRC with a fluoropyrimidine-based chemotherapy regimen containing either oxaliplatin or irinotecan, and radiographically documented progression of disease on or after treatment.

Exclusion Criteria:

* Prior treatment with a therapy targeting KRAS G12C mutation (e.g., AMG 510).
* Prior treatment with an anti-EGFR antibody (e.g., cetuximab or panitumumab).
* Active brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 30 months
  Defined as time from date of randomization to date of death due to any cause.
Progression-free Survival (PFS) | 30 months
  Defined as time from randomization until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events | 30 months
  Defined as number of patients with treatment emergent AEs.
Objective Response Rate (ORR) | 30 months
  Defined as the percent of patients documented to have a confirmed CR or PR.
Duration of Response (DOR) | 30 months
  Defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Patient Reported Outcomes (PROs) | 30 months
  To be assessed by European Quality of Life Questionnaire for Cancer Patients (QLQ-C30).
Quality of Life Assessment | 30 months
  To be assessed by European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L).

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (419):
- United States (185):
  - Local Institution - 010-855-E, Alabaster, Alabama
  - Local Institution - 010-855-B, Bessemer, Alabama
  - Local Institution - 010-855-D, Birmingham, Alabama
  - Local Institution - 010-855-A, Birmingham, Alabama
  - Local Institution - 010-855-F, Birmingham, Alabama
  - Local Institution - 010-855-C, Birmingham, Alabama
  - Local Institution - 010-855, Birmingham, Alabama
  - Local Institution - 010-996, Gilbert, Arizona
  - Local Institution - 010-566, Goodyear, Arizona
  - Local Institution - 010-989, Phoenix, Arizona
  - Local Institution - 010-978, Springdale, Arkansas
  - Local Institution - 010-573, Bakersfield, California
  - Local Institution - 010-979C, Chula Vista, California
  - Local Institution - 010-980, Fresno, California
  - Local Institution - 010-851, Fullerton, California
  - Local Institution - 010-979A, La Mesa, California
  - Local Institution - 010-958A, Los Angeles, California
  - Local Institution - 010-958, Los Angeles, California
  - Local Institution - 010-551, Los Angeles, California
  - Local Institution - 010-847, Newport Beach, California
  - Local Institution - 010-563, Redlands, California
  - Local Institution - 010-979B, San Diego, California
  - Local Institution - 010-979D, San Diego, California
  - Local Institution - 010-979, San Diego, California
  - Local Institution - 010-982, San Francisco, California
  - Local Institution - 010-561, Santa Monica, California
  - Local Institution - 010-571, Sylmar, California
  - Local Institution - 010-574, Torrance, California
  - Local Institution - 010-570, Whittier, California
  - Local Institution - 010-872-H, Aurora, Colorado
  - Local Institution - 010-810, Aurora, Colorado
  - Local Institution - 010-872-A, Boulder, Colorado
  - Local Institution - 010-872-E, Centennial, Colorado
  - Local Institution - 010-872-C, Colorado Springs, Colorado
  - Local Institution - 010-872, Denver, Colorado
  - Local Institution - 010-872-B, Denver, Colorado
  - Local Institution - 010-872-J, Lakewood, Colorado
  - Local Institution - 010-872-F, Littleton, Colorado
  - Local Institution - 010-872-G, Longmont, Colorado
  - Local Institution - 010-872-I, Pueblo, Colorado
  - Local Institution - 010-872-D, Thornton, Colorado
  - Local Institution - 010-949, Norwich, Connecticut
  - Local Institution - 010-922-A, Bonita Springs, Florida
  - Local Institution - 010-922-D, Bradenton, Florida
  - Local Institution - 010-922-E, Cape Coral, Florida
  - Local Institution - 010-922, Fort Myers, Florida
  - Local Institution - 010-922-B, Fort Myers, Florida
  - Local Institution - 010-922-C, Fort Myers, Florida
  - Local Institution - 010-984-B, Holiday, Florida
  - Local Institution - 010-829, Jacksonville, Florida
  - Local Institution - 010-923-A, Largo, Florida
  - Local Institution - 010-923-B, Largo, Florida
  - Local Institution - 010-923-C, Largo, Florida
  - Local Institution - 010-923-D, Largo, Florida
  - Local Institution - 010-923-E, Largo, Florida
  - Local Institution - 010-923-F, Largo, Florida
  - Local Institution - 010-923-G, Largo, Florida
  - Local Institution - 010-923-H, Largo, Florida
  - Local Institution - 010-923-I, Largo, Florida
  - Local Institution - 010-923-J, Largo, Florida
  - Local Institution - 010-923-K, Largo, Florida
  - Local Institution - 010-923-L, Largo, Florida
  - Local Institution - 010-923-M, Largo, Florida
  - Local Institution - 010-923-N, Largo, Florida
  - Local Institution - 010-923-O, Largo, Florida
  - Local Institution - 010-923-P, Largo, Florida
  - Local Institution - 010-990, Miami, Florida
  - Local Institution - 010-922-F, Naples, Florida
  - Local Institution - 010-922-G, Naples, Florida
  - Local Institution - 010-538, Ocala, Florida
  - Local Institution - 010-896, Orlando, Florida
  - Local Institution - 010-988, Orlando, Florida
  - Local Institution - 010-922-H, Port Charlotte, Florida
  - Local Institution - 010-923, St. Petersburg, Florida
  - Local Institution - 010-984, St. Petersburg, Florida
  - Local Institution - 010-924, Tallahassee, Florida
  - Local Institution - 010-984-A, Trinity, Florida
  - Local Institution - 010-926, West Palm Beach, Florida
  - Local Institution - 010-537, Weston, Florida
  - Local Institution - 010-956, Atlanta, Georgia
  - Local Institution - 010-986, Newnan, Georgia
  - Local Institution - 010-963, Naperville, Illinois
  - Local Institution - 010-994, Zion, Illinois
  - Local Institution - 010-569-A, Indianapolis, Indiana
  - Local Institution - 010-569, Indianapolis, Indiana
  - Local Institution - 010-991, Iowa City, Iowa
  - Local Institution - 010-920, Baton Rouge, Louisiana
  - Local Institution - 010-534, Baltimore, Maryland
  - Local Institution - 010-997, Boston, Massachusetts
  - Local Institution - 010-531A, Brownstown, Michigan
  - Local Institution - 010-531C, Dearborn, Michigan
  - Local Institution - 010-531, Detroit, Michigan
  - Local Institution - 010-531B, Novi, Michigan
  - Local Institution - 010-875, Minneapolis, Minnesota
  - Local Institution - 010-830, Rochester, Minnesota
  - Local Institution - 010-838, Saint Louis Park, Minnesota
  - Local Institution - 010-838A, Saint Louis Park, Minnesota
  - Local Institution - 010-838B, Saint Louis Park, Minnesota
  - Local Institution - 010-838C, Saint Louis Park, Minnesota
  - Local Institution - 010-838D, Saint Louis Park, Minnesota
  - Local Institution - 010-838E, Saint Louis Park, Minnesota
  - Local Institution - 010-838F, Saint Louis Park, Minnesota
  - Local Institution - 010-838G, Saint Louis Park, Minnesota
  - Local Institution - 010-838H, Saint Louis Park, Minnesota
  - Local Institution - 010-838I, Saint Louis Park, Minnesota
  - Local Institution - 010-838J, Saint Louis Park, Minnesota
  - Local Institution - 010-838K, Saint Louis Park, Minnesota
  - Local Institution - 010-838L, Saint Louis Park, Minnesota
  - Local Institution - 010-838M, Saint Louis Park, Minnesota
  - Local Institution - 010-541, Springfield, Missouri
  - Local Institution - 010-564, Lincoln, Nebraska
  - Local Institution - 010-590, Omaha, Nebraska
  - Local Institution - 010-860 - A, Henderson, Nevada
  - Local Institution - 010-860-F, Henderson, Nevada
  - Local Institution - 010-860-B, Henderson, Nevada
  - Local Institution - 010-860-D, Las Vegas, Nevada
  - Local Institution - 010-860-C, Las Vegas, Nevada
  - Local Institution - 010-860-E, Las Vegas, Nevada
  - Local Institution - 010-860, Las Vegas, Nevada
  - Local Institution - 010-918 - B, Basking Ridge, New Jersey
  - Local Institution - 010-993, Belleville, New Jersey
  - Local Institution - 010-975, East Brunswick, New Jersey
  - Local Institution - 010-992, Florham Park, New Jersey
  - Local Institution - 010-918 - D, Middletown, New Jersey
  - Local Institution - 010-918 - C, Montvale, New Jersey
  - Local Institution - 010-957, New Brunswick, New Jersey
  - Local Institution - 010-535 - D, Babylon, New York
  - Local Institution - 010-918 - A, Commack, New York
  - Local Institution - 010-918 - F, Harrison, New York
  - Local Institution - 010-813, New York, New York
  - Local Institution - 010-535 - G, New York, New York
  - Local Institution - 010-998, New York, New York
  - Local Institution - 010-918, New York, New York
  - Local Institution - 010-535 - C, Patchogue, New York
  - Local Institution - 010-535 - A, Port Jefferson, New York
  - Local Institution - 010-535 - B, Port Jefferson Station, New York
  - Local Institution - 010-535 - F, Riverhead, New York
  - Local Institution - 010-535, Shirley, New York
  - Local Institution - 010-535 - E, The Bronx, New York
  - Local Institution - 010-918 - E, Uniondale, New York
  - Local Institution - 010-585-B, Clinton, North Carolina
  - Local Institution - 010-585, Goldsboro, North Carolina
  - Local Institution - 010-585-A, Jacksonville, North Carolina
  - Local Institution - 010-893, Cincinnati, Ohio
  - Local Institution - 010-532, Oklahoma City, Oklahoma
  - Local Institution - 010-549, Oklahoma City, Oklahoma
  - Local Institution - 010-584, Tulsa, Oklahoma
  - Local Institution - 010-596, Pittsburgh, Pennsylvania
  - Local Institution - 010-981, Greenville, South Carolina
  - Local Institution - 010-921, Chattanooga, Tennessee
  - Local Institution - 010-801, Nashville, Tennessee
  - Local Institution - 010-572, Dallas, Texas
  - Local Institution - 010-879, Dallas, Texas
  - Local Institution - 010-577-B, Houston, Texas
  - Local Institution - 010-577-A, Houston, Texas
  - Local Institution - 010-577, Houston, Texas
  - Local Institution - 010-848, Houston, Texas
  - Local Institution - 010-977, Houston, Texas
  - Local Institution - 010-999, Irving, Texas
  - Local Institution - 010-878-B, Longview, Texas
  - Local Institution - 010-862, San Antonio, Texas
  - Local Institution - 010-964, Temple, Texas
  - Local Institution - 010-878, Tyler, Texas
  - Local Institution - 010-976-F, American Fork, Utah
  - Local Institution - 010-976-C, Bountiful, Utah
  - Local Institution - 010-976-D, Layton, Utah
  - Local Institution - 010-976-A, Murray, Utah
  - Local Institution - 010-976-H, Ogden, Utah
  - Local Institution - 010-976-G, Provo, Utah
  - Local Institution - 010-976-B, Salt Lake City, Utah
  - Local Institution - 010-976, Salt Lake City, Utah
  - Local Institution - 010-976-E, West Jordan, Utah
  - Local Institution - 010-919, Fairfax, Virginia
  - Local Institution - 010-597, Fredericksburg, Virginia
  - Local Institution - 010-539, Richmond, Virginia
  - Local Institution - 010-536, Richmond, Virginia
  - Local Institution - 010-533 A, Auburn, Washington
  - Local Institution - 010-576, Everett, Washington
  - Local Institution - 010-533 B, Gig Harbor, Washington
  - Local Institution - 010-533 C, Puyallup, Washington
  - Local Institution - 010-824, Seattle, Washington
  - Local Institution - 010-533, Tacoma, Washington
  - Local Institution - 010-885, Vancouver, Washington
  - Local Institution - 010-575, Morgantown, West Virginia
  - Local Institution - 010-947, Milwaukee, Wisconsin
- Argentina (6):
  - Local Institution - 010-434, Buenos Aires
  - Local Institution - 010-431, Buenos Aires
  - Local Institution - 010-432, CABA
  - Local Institution - 010-430, La Rioja
  - Local Institution - 010-448, Porto Alegre
  - Local Institution - 010-433, Viedma
- Australia (6):
  - Local Institution - 010-005, Bedford Park
  - Local Institution - 010-004, Clayton
  - Local Institution - 010-006, Garran
  - Local Institution - 010-015, Heidelberg
  - Local Institution - 010-012, Melbourne
  - Local Institution - 010-002, Waratah
- Austria (3):
  - Local Institution - 010-145, Innsbruck
  - Local Institution - 010-144, Vienna
  - Local Institution - 010-143, Wiener Neustadt
- Belgium (4):
  - Local Institution - 010-154, Brussels
  - Local Institution - 010-157, Edegem
  - Local Institution - 010-156, Ghent
  - Local Institution - 010-150, Yvoir
- Brazil (10):
  - Local Institution - 010-446, Ijuí, Rio Grande do Sul
  - Local Institution - 010-443, Porto Alegre, Rio Grande do Sul
  - Local Institution - 010-450, Blumenau, Santa Catarina
  - Local Institution - 010-442, Curitiba
  - Local Institution - 010-449, Liberdade
  - Local Institution - 010-444, Santo André
  - Local Institution - 010-440, São José do Rio Preto
  - Local Institution - 010-441, São Paulo
  - Local Institution - 010-445, São Paulo
  - Local Institution - 010-447, São Paulo
- Canada (4):
  - Local Institution - 010-481, Ottawa, Ontario
  - Local Institution - 010-483, Toronto, Ontario
  - Local Institution - 010-482, Toronto, Ontario
  - Local Institution - 010-487, Montreal, Quebec
- China (33):
  - Local Institution - 010-712, Bengbu, Anhui
  - Local Institution - 010-026, Hefei, Anhui
  - Local Institution - 010-022, Hefei, Anhui
  - Local Institution - 010-711, Hefei, Anhui
  - Local Institution - 010-717, Beijing, Beijing Municipality
  - Local Institution - 010-029, Fuzhou, Fujian
  - Local Institution - 010-031, Guangzhou, Guangdong
  - Local Institution - 010-713, Shenzhen, Guangdong
  - Local Institution - 010-715, Nanning, Guangxi
  - Local Institution - 010-021, Zhengzhou, Henan
  - Local Institution - 010-703, Wuhan, Hubei
  - Local Institution - 010-701, Wuhan, Hubei
  - Local Institution - 010-035, Changsha, Hunan
  - Local Institution - 010-714, Jiangyin, Jiangsu
  - Local Institution - 010-704, Nanjing, Jiangsu
  - Local Institution - 010-706, Nanchang, Jiangxi
  - Local Institution - 010-030, Changchun, Jilin
  - Local Institution - 010-718, Changchun, Jilin
  - Local Institution - 010-709, Shenyang, Liaoning
  - Local Institution - 010-705, Shenyang, Liaoning
  - Local Institution - 010-036, Jinan, Shandong
  - Local Institution - 010-038, Shanghai, Shanghai Municipality
  - Local Institution - 010-020, Shanghai, Shanghai Municipality
  - Local Institution - 010-708, Shanghai, Shanghai Municipality
  - Local Institution - 010-025, Shanghai Shi, Shanghai Municipality
  - Local Institution - 010-024, Shanghaishi, Shanghai Municipality
  - Local Institution - 010-710, Chengdu, Sichuan
  - Local Institution - 010-716, Neijiang, Sichuan
  - Local Institution - 010-027, Tianjin, Tianjin Municipality
  - Local Institution - 010-707, Hangzhou, Zhejiang
  - Local Institution - 010-034, Hangzhou, Zhejiang
  - Local Institution - 010-032, Hangzhou
  - Local Institution - 010-033, Hongkou Qu
- Colombia (4):
  - Local Institution - 010-460, Barranquilla
  - Local Institution - 010-462, Bogotá
  - Local Institution - 010-465, Floridablanca
  - Local Institution - 010-463, Medellín
- Czechia (4):
  - Local Institution - 010-165, Brno
  - Local Institution - 010-160, Brno
  - Local Institution - 010-162, Olomouc
  - Local Institution - 010-161, Prague
- Denmark (3):
  - Local Institution - 010-171, Copenhagen
  - Local Institution - 010-172, Odense
  - Local Institution - 010-170, Vejle
- Finland (3):
  - Local Institution - 010-180, Helsinki
  - Local Institution - 010-182, Tampere
  - Local Institution - 010-181, Turku
- France (18):
  - Local Institution - 010-209-A, Chambray-lès-Tours, Centre-Val de Loire
  - Local Institution - 010-668, Avignon
  - Local Institution - 010-208, Besançon
  - Local Institution - 010-669, Bordeaux
  - Local Institution - 010-194, Brest
  - Local Institution - 010-192, Dijon
  - Local Institution - 010-662, Lille
  - Local Institution - 010-205, Lyon
  - Local Institution - 010-682, Marseille
  - Local Institution - 010-207, Paris
  - Local Institution - 010-203, Paris
  - Local Institution - 010-204, Paris
  - Local Institution - 010-661, Paris
  - Local Institution - 010-660, Pessac
  - Local Institution - 010-667, Suresnes
  - Local Institution - 010-680, Toulouse
  - Local Institution - 010-209, Tours
  - Local Institution - 010-202, Villejuif
- Germany (12):
  - Local Institution - 010-675, Amberg
  - Local Institution - 010-657, Berlin
  - Local Institution - 010-655, Bochum
  - Local Institution - 010-227, Dresden
  - Local Institution - 010-229, Frankfurt am Main
  - Local Institution - 010-656, Hamburg
  - Local Institution - 010-658, Herne
  - Local Institution - 010-228, Mönchengladbach
  - Local Institution - 010-650, München
  - Local Institution - 010-226, München
  - Local Institution - 010-652, Reutlingen
  - Local Institution - 010-676, Ulm
- Greece (6):
  - Local Institution - 010-501, Athens
  - Local Institution - 010-232, Cholargós
  - Local Institution - 010-238, Heraklion
  - Local Institution - 010-235, Larissa
  - Local Institution - 010-231, Thessaloniki
  - Local Institution - 010-230, Thessaloniki
- Hong Kong (2):
  - Local Institution - 010-048, Central
  - Local Institution - 010-046, Hong Kong
- Ireland (5):
  - Local Institution - 010-250, Dublin
  - Local Institution - 010-252, Dublin
  - Local Institution - 010-253, Dublin
  - Local Institution - 010-254, Dublin
  - Local Institution - 010-251, Dublin
- Italy (14):
  - Local Institution - 010-292, Avellino
  - Local Institution - 010-290, Biella
  - Local Institution - 010-299, Cagliari
  - Local Institution - 010-286, Candiolo
  - Local Institution - 010-287, Lido di Camaiore
  - Local Institution - 010-270, Meldola
  - Local Institution - 010-278, Milan
  - Local Institution - 010-293, Milan
  - Local Institution - 010-271, Napoli
  - Local Institution - 010-297, Padua
  - Local Institution - 010-294, Pisa
  - Local Institution - 010-291, Reggio Emilia
  - Local Institution - 010-295, Roma
  - Local Institution - 010-289, Torino
- Malaysia (6):
  - Local Institution - 010-070, Johor Bahru, Johor
  - Local Institution - 010-077, Kota Kinabalu, Sabah
  - Local Institution - 010-071, Petaling Jaya, Selangor
  - Local Institution - 010-073, Kuala Lumpur
  - Local Institution - 010-074, Kuala Lumpur
  - Local Institution - 010-072, Putrajaya
- Mexico (7):
  - Local Institution - 010-474, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 010-472, Guadalajara, Jalisco
  - Local Institution - 010-477, Guadalajara, Jalisco
  - Local Institution - 010-473, Mexico City, Mexico City
  - Local Institution - 010-476, Cuernavaca, Morelos
  - Local Institution - 010-475, San Juan del Río, Querétaro
  - Local Institution - 010-471, Colonia Centro Orizaba, Veracruz
- Netherlands (4):
  - Local Institution - 010-632, Amsterdam
  - Local Institution - 010-306, Amsterdam
  - Local Institution - 010-630, Nijmegen
  - Local Institution - 010-307, Utrecht
- Poland (4):
  - Local Institution - 010-328, Gdansk
  - Local Institution - 010-327, Otwock
  - Local Institution - 010-322, Warsaw
  - Local Institution - 010-787, Warsaw
- Portugal (5):
  - Local Institution - 010-332, Braga
  - Local Institution - 010-337, Lisbon
  - Local Institution - 010-640, Lisbon
  - Local Institution - 010-331, Porto
  - Local Institution - 010-339, Porto
- Puerto Rico (3):
  - Local Institution - 010-902, San Juan
  - Local Institution - 010-903, San Juan
  - Local Institution - 010-900, San Juan
- Romania (8):
  - Local Institution - 010-347, Baia Mare
  - Local Institution - 010-349, Brasov
  - Local Institution - 010-512, Bucharest
  - Local Institution - 010-344, Cluj-Napoca
  - Local Institution - 010-340, Cluj-Napoca
  - Local Institution - 010-343, Craiova
  - Local Institution - 010-511, Ovidiu
  - Local Institution - 010-510, Timișoara
- Singapore (5):
  - Local Institution - 010-090, Singapore
  - Local Institution - 010-093, Singapore
  - Local Institution - 010-095, Singapore
  - Local Institution - 010-092, Singapore
  - Local Institution - 010-091, Singapore
- South Korea (15):
  - Local Institution - 010-116, Anyang-si
  - Local Institution - 010-111, Busan
  - Local Institution - 010-119, Busan
  - Local Institution - 010-525, Daejeon
  - Local Institution - 010-117, Goyang-si
  - Local Institution - 010-100, Hwasun-gun
  - Local Institution - 010-520, Seongnam-si
  - Local Institution - 010-105, Seoul
  - Local Institution - 010-108, Seoul
  - Local Institution - 010-118, Seoul
  - Local Institution - 010-104, Seoul
  - Local Institution - 010-114, Seoul
  - Local Institution - 010-109, Seoul
  - Local Institution - 010-115, Suwon
  - Local Institution - 010-524, Yangsan
- Spain (15):
  - Local Institution - 010-613, A Coruña
  - Local Institution - 010-610, Badalona
  - Local Institution - 010-612, Barcelona
  - Local Institution - 010-600, Barcelona
  - Local Institution - 010-621, Córdoba
  - Local Institution - 010-620, LHospitalet de Llobregat
  - Local Institution - 010-619, Madrid
  - Local Institution - 010-601, Madrid
  - Local Institution - 010-617, Madrid
  - Local Institution - 010-624, Madrid
  - Local Institution - 010-623, Pamplona
  - Local Institution - 010-622, Sabadell
  - Local Institution - 010-604, Santander
  - Local Institution - 010-618, Valencia
  - Local Institution - 010-625, Valencia
- Taiwan (7):
  - Local Institution - 010-129, Changhua
  - Local Institution - 010-121, Kaohsiung City
  - Local Institution - 010-124, Taichung
  - Local Institution - 010-122, Tainan
  - Local Institution - 010-123, Tainan
  - Local Institution - 010-120, Taipei
  - Local Institution - 010-125, Taoyuan District
- Thailand (5):
  - Local Institution - 010-132, Bang Phlat
  - Local Institution - 010-134, Bangkok
  - Local Institution - 010-131, Chiang Mai
  - Local Institution - 010-130, Hat Yai
  - Local Institution - 010-133, Khlong Toey
- Local Institution - 010-424, Sumy, Ukraine
- United Kingdom (12):
  - Local Institution - 010-412, Aberdeen
  - Local Institution - 010-410, Birmingham
  - Local Institution - 010-413, Cambridge
  - Local Institution - 010-411, Dorset
  - Local Institution - 010-400, Glasgow
  - Local Institution - 010-403, Kent
  - Local Institution - 010-414, Leeds
  - Local Institution - 010-402, London
  - Local Institution - 010-405, London
  - Local Institution - 010-406, London
  - Local Institution - 010-407, Manchester
  - Local Institution - 010-404, Middlesex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com